CLINICAL TRIAL: NCT02768415
Title: Phase II Study of Apatinib Combined With Oral Vinorelbine in Pretreated Metastatic HER2 Negative Breast Cancer
Brief Title: Study of Apatinib Combined With Oral Vinorelbine in Metastatic HER2 Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-046
Record Dates: First submitted 2016-05-04; First posted 2016-05-11 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib; Vinorelbine

ARMS (1):
- lapatinib+oral vinorelbine (Experimental): apatinib 425/500mg qd, 21days/cycle
  oral vinorelbine 60mg/m2 d1, 8, 15 21days/cycle*3cycles, after 3 cycles: 80mg/m2 d1, 8, 15 21days/cycle
  Interventions: Drug: Apatinib; Drug: Oral Vinorelbine

INTERVENTIONS:
Drug: Apatinib
Drug: Oral Vinorelbine

SUMMARY:
The hypothesis of this study is to discover if the all-oral therapy with apatinib plus oral vinorelbine can shrink or slow the growth of pretreated HER2 negative metastatic breast cancer.

DETAILED DESCRIPTION:
Apatinib is an orally administered second-generation blocker of the phosphorylation of the tyrosine residues within the intracellular domain of VEGF receptor 2 (VEGFR2). A prospective, open label, phase II multicenter trial of apatinib in heavily pretreated patients with metastatic triple-negative breast cancer demonstrated that the daily dose of apatinib 500 mg/day is active in pretreated metastatic TNBC with encouraging rates of disease stabilization and PFS.

Vinorelbine is a highly active drug in the treatment of MBC, both as a single agent or in combination regimens, and is well tolerated, with a low incidence of severe toxicity. Clinical trials demonstrated oral NVB provided comparable effectiveness to iv NVB. and oral availability allows using different schedules.

The NCCN guideline introduces that combination chemotherapy is one of the standard treatment options in metastatic breast cancer, especially in patients with visceral metastases and/or need of rapid symptom or disease control.

Theoretically, anti-angiogenesis regimen combined with chemotherapy may present increasing therapeutic effect. Related researches are urgently needed to find optimal combined therapy.

The hypothesis of this study is to discover if the all-oral therapy with apatinib plus oral vinorelbine can shrink or slow the growth of pretreated HER2 negative breast cancer. The safety of the combination will also be studied. Patients physical state, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if this combination is safe and effective in pretreated HER2 negative metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 year-old women; HER2 negative(immunohistochemistry or fluorescence in situ hybridization);
2. ECOG score: 0-1, expected survival time ≥ 3months;
3. Pathologically or cytologically confirmed breast cancer;
4. Anthracycline- / taxane- pretreated (adjuvant, neoadjuvant) breast cancer patients who have failed from 1-2 standard chemotherapies after recurrence and metastasis;
5. According to RECIST 1.1, exist at least ≥1 measurable lesion(CT >1cm，other examination >2cm) ;
6. The patients have enough organ function. The laboratory test indexes must comply with the following requirements:

   Blood routine: neutrophil≥1.5G/L, platelet count ≥80G/L, hemoglobin ≥90g/L Liver function: serum bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST≤2.5 times the upper limit of normal value; ALT and AST≤5 times the upper limit of normal value when liver metastasis Renal function: serum creatinine ≤ 1.0times the upper limit of normal value, creatinine clearance >50ml/min（Cockcroft-Gault formula)
7. Women of child-bearing age should be carried out pregnancy test (serum or urine) within 7 days before recruit, the results should be negative; and are willing to adopt the appropriate methods of contraception during the trial and 8 weeks after last administration；
8. Can swallow oral drugs;
9. The patients have good compliance to the therapy and follow-up to be scheduled and are able to understand the study protocol and sign the Informed Consent Form.

Exclusion Criteria:

1. The patients in pregnancy or lactation growth period and did not take effective contraception;
2. The patients who received ≥3 chemotherapies（Do not include endocrine therapy）after recurrence and metastasis; involved in other clinical trials four weeks prior to the start of the study;
3. The patients with a variety of factors that affect the oral administration and absorption of drugs；
4. The patients previously received anti-VEFG of anti-VEGFR therapies；
5. The patients with rapid progression of viscera invasion(liver lesion >1/2 viscera area or liver dysfunction);
6. The patients have uncontrollable mental illness.
7. The patients who had serious adverse effect to oral vinorelbine or were allergic to vinorelbine.
8. The patients who have only bone metastasis without other measurable lesion;
9. The patients experience severe cardiovascular diseases;
10. The patients experience severe upper gastrointestinal ulcer or malabsorption syndrome.
11. Abnormal bone marrow functions(neutrophil<1.5G/L, platelet count <75G/L, hemoglobin <90g/L)；
12. Abnormal renal function(serum creatinine > 1.5 times the upper limit of normal value)；
13. Abnormal liver function(serum bilirubin ≤ 1.5 times the upper limit of normal value);
14. The patients have uncontrollable brain metastasis;
15. The patients do not have good compliance to the therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) among metastatic HER2 negative breast cancer treated with apatinib and oral vinorelbine | up to 1 year after the last patient enrolled

SECONDARY OUTCOMES:
remission rate (RR) among metastatic HER2 negative breast cancer treated with apatinib and oral vinorelbine | up to 1 year after the last patient enrolled
overall survival (OS) among metastatic HER2 negative breast cancer treated with apatinib and oral vinorelbine | up to 1 year after the last patient enrolled
overall response rate (ORR) among metastatic HER2 negative breast cancer treated with apatinib and oral vinorelbine | up to 1 year after the last patient enrolled
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 1 year after the last patient enrolled
Potential biomarkers to predict efficacy, drug resistance and side effects of anti-angiogenic therapy plus chemotherapy in advanced breast cancer. | up to 1 year after the last patient enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China